CLINICAL TRIAL: NCT01880814
Title: Using SMART Experimental Design to Personalize Treatment for Child Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dikla Eckshtain, PhD, Instructor in Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5K23MH093491 (NIH)
Record Dates: First submitted 2013-06-10; First posted 2013-06-19 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2020-08

CONDITIONS: Depression
Keywords: Depression, child, CBT, parent training, personalized treatment
MeSH Terms: conditions — Depression; Color Vision Defects | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (CBT) (Experimental): Type of talk therapy that focuses on individual behavioral and cognitive skills.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Caregiver-Child Treatment (Experimental): Type of talk therapy that involves the child and the caregiver and focuses on behavioral and cognitive skills.
  Interventions: Behavioral: Caregiver-Child Treatment

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Children will first be randomized into Stage 1 of CBT or Caregiver-Child Treatment. Stage 1 will include six sessions. After Stage 1, child's response to treatment will be evaluated. Responders will be re-randomized into Stage 2 of no treatment or continuation of CBT. If randomized to no treatment, termination session will be completed. If randomized to continuation of CBT, the treatment will include six sessions and a termination session. Insufficient responders will be re-randomized into Stage 2 of continuation of CBT or Caregiver-Child Treatment. Stage 2 will include six sessions and a termination session.
  Arms: Cognitive Behavioral Therapy (CBT)
Behavioral: Caregiver-Child Treatment — Children will first be randomized into Stage 1 of CBT or Caregiver-Child Treatment. Stage 1 will include six sessions. After Stage 1, child's response to treatment will be evaluated. Responders will be re-randomized into Stage 2 of no treatment or continuation of Caregiver-Child Treatment. If randomized to no treatment, termination session will be completed. If randomized to continuation of Caregiver-Child Treatment, the treatment will include six sessions and a termination session. Insufficient responders will be re-randomized into Stage 2 of continuation of Caregiver-Child Treatment or CBT. Stage 2 will include six sessions and a termination session.
  Arms: Caregiver-Child Treatment

SUMMARY:
The purpose of the study is:

1. To conduct a pilot SMART (Sequential, Multiple Assignment, Randomized) study with the long-term goal of developing a personalized treatment for child depression.
2. To collect pilot data on ways to personalize treatment for child depression using cognitive behavioral therapy (CBT), caregiver-child treatment, or both.

DETAILED DESCRIPTION:
Child depression is among the most prevalent and impairing pediatric conditions and constitutes a major public health concern. Unfortunately, treatment benefits are relatively modest and short-lived with sizeable percentages of children who maintain depressive symptoms following treatment. This problem may be addressed in part by personalizing treatment, including determining which children will benefit from CBT, which children will benefit from caregiver-child treatment, and which children will benefit from both. The goal of the current study is to pilot test an innovative experimental design called Sequential, Multiple Assignment, Randomized Trial (SMART), which is used for development of personalized treatments, collect pilot data, and assess the acceptability and feasibility of using this design, in preparation for a full-scale SMART in a larger clinical trial and for the development of personalized treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Current diagnosis of Major Depressive Disorder (MDD), Dysthymic Disorder (DD), or Depressive Disorder Not Otherwise Specified (NOS).
2. If receiving psychiatric medication, dose should be stable for at least three months at enrollment.

Exclusion Criteria:

1. A disorder other than depression as primary diagnosis.
2. Autism Spectrum Disorders and Pervasive Developmental Delay or Disorder.
3. Mental Retardation.
4. Psychotic Disorders and Schizophrenia.
5. Mania or Hypomania disorders.
6. Acute suicidal behavior and/or acute plan that require higher level of care, and being hospitalized over the past year for a suicide attempt or for threatening to commit suicide.
7. Participation in additional psychotherapy.
8. Caregiver and/or children do not speak English.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2013-06; Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Schedule for Affective Disorders and Schizophrenia for School-Aged Children-Present and Lifetime Versions (K-SADS-PL) | Pre-treatment, Stage 1, Stage 2, 3-month follow-up
  Clinician-administered semi-structured interview with children and caregivers assessing present episode and lifetime history of psychiatric diagnoses based on DSM-IV criteria.
Children's Depression Rating Scale-Revised (CDRS-R) | Pre-treatment, Stage 1, Stage 2, 3-month follow-up
  Clinician-administered semi-structured child interview of depression.
Children's Depression Inventory 2: Self Report (CDI2:SR) | Pre-treatment, Stage 1, Stage 2, 3-month follow-up
  Child self-report questionnaire assessing depressive symptoms.
Children's Depression Inventory 2:Parent (CDI2:P) | Pre-treatment, Stage 1, Stage 2, 3-month follow-up, before each session
  Parent-report questionnaire assessing child's depressive symptoms.
Clinical Global Impression (CGI) | Pre-treatment, Stage 1, Stage 2, 3-month follow-up
  Clinician assessment of child's symptom severity and level of improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States